CLINICAL TRIAL: NCT01107275
Title: Compare Immunogenicity, Safety and Long-term Booster Response After Primary Vaccination With 2 Intradermal Doses Versus 3 Intradermal Doses of PCEC Rabies Vaccine (Rabipur) in Healthy School Children in Thailand (5-8 Years of Age)
Brief Title: Early Rabies Vaccine Immunization in Primary School Children
Acronym: I49P1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Provincial Public Health Office, Phetchabun (Other Government)
Responsible Party: Thavatchai Kamoltham, Ministry of health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: I49P1
Record Dates: First submitted 2010-04-16; First posted 2010-04-20 (Estimated); Last update posted 2010-04-20 (Estimated); Status verified 2010-04

CONDITIONS: Rabies Prevention
Keywords: Rabies; PCECV; pre-exposure immunization; intradermal; children
MeSH Terms: conditions — Rabies | interventions — Rabies Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 primary ID doses (Experimental): two doses of rabies vaccines given intradermally on days 0 and 28
  Interventions: Biological: rabies vaccine
- 3 primary ID doses (Experimental): three doses of rabies vaccines given intradermally on days 0, 7, and 28
  Interventions: Biological: rabies vaccine

INTERVENTIONS:
Biological: rabies vaccine — intradermal vaccination
  Other Names: PCECV, Rabipur

SUMMARY:
700 male and female healthy school-children (age 5 to 8) in Thailand were randomized to receive 2 or 3 primary rabies vaccine doses (PCECV, Rabipur) given intradermally in a dose of 0.1mL into the skin in the deltoid region. In a subset of 100 children blood was taken for rabies virus neutralizing antibody determination on day 49. All subjects were randomized to receive 2 booster doses (the recommended vaccination schedule for pre-immunized individuals in case of an exposure) on days 0 and 3, one, three or five years later. Blood was taken before and after booster for up to one year.Safety and tolerability of the vaccine was assessed and persistence of immune response up to 1 year after the booster doses.

ELIGIBILITY:
Inclusion criteria:

Male and female 5-8 years old school children will be included in the study if:

* Their parents or legal guardians have given the written informed consent prior to study entry;
* They are in good health at time of study entry as determined by medical history, physical examination and clinical judgment of the investigator;
* They are available for all the visits scheduled in the study.

Exclusion criteria:

Subjects are not to be enrolled into the study if:

* They have a history of rabies immunization;
* They have an acute infectious disease at the time of study entry;
* They are under treatment with parenteral and/or oral steroids, immunosuppressive drugs, phenytoin or other specific anti-inflammatory drugs, or have taken chloroquine during the two month period before enrolment;
* They have a known immunodeficiency or an autoimmune disease;
* They have a known hypersensitivity to neomycin, tetracycline or amphotericin-B;
* They have planned surgery during the first study period (49 days);
* They are participating in any other trial of an investigational agent;
* They have any condition which in the opinion of the investigator, might interfere with the evaluation of the study objectives.
* The family plans to leave the area of the study site before the end of the study period.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 703 (Actual)
Dates: Start 2002-11; Primary Completion 2004-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
rabies virus neuralizing antibody, assessed by RFFIT | seven days after the first booster dose
  rabies virus neuralizing antibody concentrations were measured in serum samples using the rapid fluorescent focus inhibition test (RFFIT)

SECONDARY OUTCOMES:
rabies virus neuralizing antibody, assessed by RFFIT | one year after the first booster dose
  rabies virus neuralizing antibody concentrations were measured in serum samples using the rapid fluorescent focus inhibition test (RFFIT)
rabies virus neuralizing antibody, assessed by RFFIT | immediately before administration of the first booster dose
  rabies virus neuralizing antibody concentrations were measured in serum samples using the rapid fluorescent focus inhibition test (RFFIT)

CONTACTS AND LOCATIONS:
Overall Officials: Thavatchai Kamoltham, MD, Principal Investigator — Provincial PHO
Locations (1):
- Phetchabun Province primary schools, Phetchabun, Phetchabun, Thailand

REFERENCES:
- [Result] Kamoltham T, Thinyounyong W, Phongchamnaphai P, Phraisuwan P, Khawplod P, Banzhoff A, Malerczyk C. Pre-exposure rabies vaccination using purified chick embryo cell rabies vaccine intradermally is immunogenic and safe. J Pediatr. 2007 Aug;151(2):173-7. doi: 10.1016/j.jpeds.2007.02.044. PMID 17643772